CLINICAL TRIAL: NCT03198572
Title: Efficacy and Safety of Berberine in Non-alcoholic Steatohepatitis: a Multicentre, Randomised, Placebo-controlled Trial
Brief Title: Efficacy and Safety of Berberine in Non-alcoholic Steatohepatitis
Acronym: EASYBEinNASH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); The Affiliated Hospital of Hangzhou Normal University (Other); Tianjin Third Central Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Xinjiang Medical University (Other)
Responsible Party: Principal Investigator, Xin Gao, Director, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016ZSLC04
Record Dates: First submitted 2017-06-18; First posted 2017-06-26 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Non-alcoholic Steatohepatitis
Keywords: Non-alcoholic steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Berberine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Berberine (Experimental): Berberine was taken orally 0.5g three times per day for 48 weeks, based on lifestyle intervention.
  Interventions: Behavioral: Lifestyle intervention; Drug: Berberine
- Placebo (Placebo Comparator): Placebo was taken orally 0.5g three times per day for 48 weeks, based on lifestyle intervention.
  Interventions: Behavioral: Lifestyle intervention; Drug: Placebo

INTERVENTIONS:
Behavioral: Lifestyle intervention — Lifestyle intervention is consisted of diet control and aerobic exercise. calorie restriction: to subtract 500 kcal from daily calorie intake aerobic exercise: medium intensity aerobic exercise for more than 150 min per week with heart rate around 50-70% of the maximal heart rate.
Drug: Placebo — placebo tablets 0.5 tid, 30 minutes before each meal, for 48weeks
  Arms: Placebo
Drug: Berberine — Berberine tablets 0.5 tid, 30 minutes before each meal, for 48weeks
  Arms: Berberine

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of berberine treatment on Non-alcoholic Steatohepatitis.

DETAILED DESCRIPTION:
This is a multicenter, double-blinded, randomized, placebo-controlled clinical trial to investigate the efficacy and safety of berberine on subjects with Non-alcoholic Steatohepatitis.Patients with biopsy-proven non-alcoholic steatohepatitis (NASH) from 18-65 years of age were enrolled. Patients should had no excessive alcohol intake or use of any hepatoprotective or hepatotoxicity medication within 3 months before enrollment.Patients will have an screening period 12 weeks, and a 48-week double-blinded treatment period.

ELIGIBILITY:
The inclusion criteria are as follows:

1. 18-75 years old, no limitation for ethnicity and gender.
2. BMI is no more than 40 kg/m2.
3. Patients with NASH based on liver biopsy obtained within 24 weeks before randomization. The histological evidence of NASH is defined as NAS ≥5 [] or NAS ≥4 with a minimum score of 1 for all of three components (steatosis, hepatocyte ballooning, and lobular inflammation), the diagnosis of NASH for EASYBEinNASH eligibility is based on reviews by three pathologists. If there are controversial pathologic diagnosis, at least 2 of the 3 pathologists are consistent with the pathologic diagnosis, which will be the final pathological diagnosis. If there are three different pathological diagnoses, it needs to be discussed and make a judgment by the chief pathologist to form the final pathology report.
4. For patients with impaired glucose metabolism, one of the three following conditions needs to be met.

   ① For patients diagnosed as impaired glucose regulation, they will be treated with lifestyle intervention without hypoglycemic drugs;

   ② For patients diagnosed as diabetes and treated with hypoglycemic drugs, the treatment regimen should not be changed and the dosage should remain stable for more than 2 months before randomization;

   ③ For patients diagnosed as diabetes and treated with lifestyle intervention without hypoglycemic drugs, the treatment regimen should not be changed before randomization.
5. All participants agree to sign the informed consent form.

Exclusion criteria

1. Excessive alcohol intake ( > 140 g per week for men and >70 g per week for women within 6 months before enrollment);
2. Liver enzymes (ALT or aspartate aminotransferase(AST) is 5 times higher than the upper limit of normal range;
3. Liver diseases caused by other reasons, such as alcohol abuse, viral hepatitis, drugs, auto-immune hepatitis, hereditary liver disease, liver cirrhosis, liver cancer, etc;
4. Biliary tract diseases, biliary obstructive disease, etc;
5. Other diseases that affect glucose and lipid metabolism, such as hypothyroidism, hyperthyroidism, hypercortisolism, etc;
6. Diabetic patients with poor blood glucose control: HbA1c >9.5%;
7. Use of drugs that may affect the outcome measures of this study 3 months before enrollment, including pioglitazone, GLP-1 receptor agonist, DPP-4 inhibitor, insulin, and glycyrrhizic acid preparation, etc;
8. Chronic kidney disease or severe renal impairment, defined as serum creatinine greater than 2.0mg/dL (176.8umol/L);
9. Life expectancy is no more than 5 years;
10. Pregnant or planning to become pregnant within the next 64 weeks for female participant;
11. Any situation that may affect the implementation or results of the study;
12. Continuous use of drugs that may affect steatohepatitis 3 months before enrollment, such as glucocorticoids, methotrexate, etc;
13. Subjects participated in other clinical trials in the past 4 weeks; The researchers did not think they were suitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-08-16 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Improvement in histologic features of nonalcoholic steatohepatitis by NAFLD activity score (NAS) | 48 weeks
  A separate system of scoring the histological features of nonalcoholic fatty liver disease (NAFLD) called the NAFLD Activity Score (NAS) was used. An improvement in histologic findings require an improvement by 1 or more points in the hepatocellular ballooning score; no increase in the fibrosis score; and either a decrease in the activity score for nonalcoholic fatty liver disease to a score of 3 or less or a decrease in the activity score of at least 2 points, with at least a 1-point decrease in either the lobular inflammation or steatosis score.

SECONDARY OUTCOMES:
Improvement in the composites of NAFLD activity scores for steatosis, lobular inflammation, hepatocellular ballooning | 48 weeks
  NAFLD activity score (NAS) is composed of steatosis (scale of 0 to 3), lobular inflammation (scale of 0 to 3), hepatocellular ballooning (scale of 0 to 2). Alteration in each component of NAS is measured.
Improvement in liver histological fibrosis staging | 48 weeks
  Fibrosis staging was measured as following criteria: 0=none, 1=perisinusoidal or periportal fibrosis, 2=perisinusoidal and portal/periportal fibrosis, 3=bridging fibrosis, and 4=cirrhosis.the definition of fibrosis stages improvement requires at least one stage.
Resolution of NASH | 48 weeks
  Resolution of NASH was defined as a diagnosis of no steatohepatitis at 48 weeks among those with possible or definite NASH at baseline.
Change in anthropometric measures | 48 weeks
  including BMI etc
Change in blood biochemistry | 48 weeks
  including serum aminotransferase levels etc
Change in liver fat content | 48 weeks
  liver fat content determined by 1H MRS (in part of clinical centers)
Change in serum cytokeratin 18 (CK-18) in U/L | 48 weeks
  serum cytokeratin 18 (CK-18) in U/L

CONTACTS AND LOCATIONS:
Overall Officials: Xin Gao, Principal Investigator — Fudan University
Locations (6):
- China (6):
  - Department of Endocrinology and Metabolism,Shanghai 6th People's Hospital, Shanghai, Shanghai Municipality
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou
  - Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Tianjin Third Central Hospital, Tianjin
  - Xinjiang Medical University, Ürümqi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Browning JD, Szczepaniak LS, Dobbins R, Nuremberg P, Horton JD, Cohen JC, Grundy SM, Hobbs HH. Prevalence of hepatic steatosis in an urban population in the United States: impact of ethnicity. Hepatology. 2004 Dec;40(6):1387-95. doi: 10.1002/hep.20466. PMID 15565570
- [Background] Williams CD, Stengel J, Asike MI, Torres DM, Shaw J, Contreras M, Landt CL, Harrison SA. Prevalence of nonalcoholic fatty liver disease and nonalcoholic steatohepatitis among a largely middle-aged population utilizing ultrasound and liver biopsy: a prospective study. Gastroenterology. 2011 Jan;140(1):124-31. doi: 10.1053/j.gastro.2010.09.038. Epub 2010 Sep 19. PMID 20858492
- [Background] Li Z, Xue J, Chen P, Chen L, Yan S, Liu L. Prevalence of nonalcoholic fatty liver disease in mainland of China: a meta-analysis of published studies. J Gastroenterol Hepatol. 2014 Jan;29(1):42-51. doi: 10.1111/jgh.12428. PMID 24219010
- [Background] Garcia-Monzon C, Martin-Perez E, Iacono OL, Fernandez-Bermejo M, Majano PL, Apolinario A, Larranaga E, Moreno-Otero R. Characterization of pathogenic and prognostic factors of nonalcoholic steatohepatitis associated with obesity. J Hepatol. 2000 Nov;33(5):716-24. doi: 10.1016/s0168-8278(00)80301-3. PMID 11097478
- [Background] Gupte P, Amarapurkar D, Agal S, Baijal R, Kulshrestha P, Pramanik S, Patel N, Madan A, Amarapurkar A, Hafeezunnisa. Non-alcoholic steatohepatitis in type 2 diabetes mellitus. J Gastroenterol Hepatol. 2004 Aug;19(8):854-8. doi: 10.1111/j.1440-1746.2004.03312.x. PMID 15242486
- [Background] Musso G, Gambino R, Cassader M, Pagano G. Meta-analysis: natural history of non-alcoholic fatty liver disease (NAFLD) and diagnostic accuracy of non-invasive tests for liver disease severity. Ann Med. 2011 Dec;43(8):617-49. doi: 10.3109/07853890.2010.518623. Epub 2010 Nov 2. PMID 21039302
- [Background] Kotronen A, Yki-Jarvinen H. Fatty liver: a novel component of the metabolic syndrome. Arterioscler Thromb Vasc Biol. 2008 Jan;28(1):27-38. doi: 10.1161/ATVBAHA.107.147538. Epub 2007 Aug 9. PMID 17690317
- [Background] Targher G, Day CP, Bonora E. Risk of cardiovascular disease in patients with nonalcoholic fatty liver disease. N Engl J Med. 2010 Sep 30;363(14):1341-50. doi: 10.1056/NEJMra0912063. No abstract available. PMID 20879883
- [Background] Cali AM, Zern TL, Taksali SE, de Oliveira AM, Dufour S, Otvos JD, Caprio S. Intrahepatic fat accumulation and alterations in lipoprotein composition in obese adolescents: a perfect proatherogenic state. Diabetes Care. 2007 Dec;30(12):3093-8. doi: 10.2337/dc07-1088. Epub 2007 Aug 23. PMID 17717283
- [Background] Shen L. Treatment implication from the potential association between nonalcoholic fatty liver disease and cardiovascular disease. Hepatology. 2011 Jul;54(1):377-8. doi: 10.1002/hep.24213. No abstract available. PMID 21710476
- [Background] Schwimmer JB, Pardee PE, Lavine JE, Blumkin AK, Cook S. Cardiovascular risk factors and the metabolic syndrome in pediatric nonalcoholic fatty liver disease. Circulation. 2008 Jul 15;118(3):277-83. doi: 10.1161/CIRCULATIONAHA.107.739920. Epub 2008 Jun 30. PMID 18591439
- [Background] Hamaguchi M, Kojima T, Takeda N, Nakagawa T, Taniguchi H, Fujii K, Omatsu T, Nakajima T, Sarui H, Shimazaki M, Kato T, Okuda J, Ida K. The metabolic syndrome as a predictor of nonalcoholic fatty liver disease. Ann Intern Med. 2005 Nov 15;143(10):722-8. doi: 10.7326/0003-4819-143-10-200511150-00009. PMID 16287793
- [Background] Lin SC, Ang B, Hernandez C, Bettencourt R, Jain R, Salotti J, Richards L, Kono Y, Bhatt A, Aryafar H, Lin GY, Valasek MA, Sirlin CB, Brouha S, Loomba R. Cardiovascular risk assessment in the treatment of nonalcoholic steatohepatitis: a secondary analysis of the MOZART trial. Therap Adv Gastroenterol. 2016 Mar;9(2):152-61. doi: 10.1177/1756283X15621232. PMID 26929777
- [Background] Marchesini G, Moscatiello S, Di Domizio S, Forlani G. Obesity-associated liver disease. J Clin Endocrinol Metab. 2008 Nov;93(11 Suppl 1):S74-80. doi: 10.1210/jc.2008-1399. PMID 18987273
- [Background] Kistler KD, Brunt EM, Clark JM, Diehl AM, Sallis JF, Schwimmer JB; NASH CRN Research Group. Physical activity recommendations, exercise intensity, and histological severity of nonalcoholic fatty liver disease. Am J Gastroenterol. 2011 Mar;106(3):460-8; quiz 469. doi: 10.1038/ajg.2010.488. Epub 2011 Jan 4. PMID 21206486
- [Background] Chalasani N, Younossi Z, Lavine JE, Diehl AM, Brunt EM, Cusi K, Charlton M, Sanyal AJ. The diagnosis and management of non-alcoholic fatty liver disease: practice Guideline by the American Association for the Study of Liver Diseases, American College of Gastroenterology, and the American Gastroenterological Association. Hepatology. 2012 Jun;55(6):2005-23. doi: 10.1002/hep.25762. No abstract available. PMID 22488764
- [Background] Eckel RH, Jakicic JM, Ard JD, de Jesus JM, Houston Miller N, Hubbard VS, Lee IM, Lichtenstein AH, Loria CM, Millen BE, Nonas CA, Sacks FM, Smith SC Jr, Svetkey LP, Wadden TA, Yanovski SZ; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2013 AHA/ACC guideline on lifestyle management to reduce cardiovascular risk: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2014 Jul 1;63(25 Pt B):2960-84. doi: 10.1016/j.jacc.2013.11.003. Epub 2013 Nov 12. No abstract available. PMID 24239922
- [Background] Musso G, Gambino R, Cassader M, Pagano G. A meta-analysis of randomized trials for the treatment of nonalcoholic fatty liver disease. Hepatology. 2010 Jul;52(1):79-104. doi: 10.1002/hep.23623. PMID 20578268
- [Background] Sanyal AJ, Chalasani N, Kowdley KV, McCullough A, Diehl AM, Bass NM, Neuschwander-Tetri BA, Lavine JE, Tonascia J, Unalp A, Van Natta M, Clark J, Brunt EM, Kleiner DE, Hoofnagle JH, Robuck PR; NASH CRN. Pioglitazone, vitamin E, or placebo for nonalcoholic steatohepatitis. N Engl J Med. 2010 May 6;362(18):1675-85. doi: 10.1056/NEJMoa0907929. Epub 2010 Apr 28. PMID 20427778
- [Background] Neuschwander-Tetri BA, Loomba R, Sanyal AJ, Lavine JE, Van Natta ML, Abdelmalek MF, Chalasani N, Dasarathy S, Diehl AM, Hameed B, Kowdley KV, McCullough A, Terrault N, Clark JM, Tonascia J, Brunt EM, Kleiner DE, Doo E; NASH Clinical Research Network. Farnesoid X nuclear receptor ligand obeticholic acid for non-cirrhotic, non-alcoholic steatohepatitis (FLINT): a multicentre, randomised, placebo-controlled trial. Lancet. 2015 Mar 14;385(9972):956-65. doi: 10.1016/S0140-6736(14)61933-4. Epub 2014 Nov 7. PMID 25468160
- [Background] Belfort R, Harrison SA, Brown K, Darland C, Finch J, Hardies J, Balas B, Gastaldelli A, Tio F, Pulcini J, Berria R, Ma JZ, Dwivedi S, Havranek R, Fincke C, DeFronzo R, Bannayan GA, Schenker S, Cusi K. A placebo-controlled trial of pioglitazone in subjects with nonalcoholic steatohepatitis. N Engl J Med. 2006 Nov 30;355(22):2297-307. doi: 10.1056/NEJMoa060326. PMID 17135584
- [Background] Armstrong MJ, Gaunt P, Aithal GP, Barton D, Hull D, Parker R, Hazlehurst JM, Guo K; LEAN trial team; Abouda G, Aldersley MA, Stocken D, Gough SC, Tomlinson JW, Brown RM, Hubscher SG, Newsome PN. Liraglutide safety and efficacy in patients with non-alcoholic steatohepatitis (LEAN): a multicentre, double-blind, randomised, placebo-controlled phase 2 study. Lancet. 2016 Feb 13;387(10019):679-690. doi: 10.1016/S0140-6736(15)00803-X. Epub 2015 Nov 20. PMID 26608256
- [Background] Zhang Y, Li X, Zou D, Liu W, Yang J, Zhu N, Huo L, Wang M, Hong J, Wu P, Ren G, Ning G. Treatment of type 2 diabetes and dyslipidemia with the natural plant alkaloid berberine. J Clin Endocrinol Metab. 2008 Jul;93(7):2559-65. doi: 10.1210/jc.2007-2404. Epub 2008 Apr 8. PMID 18397984
- [Background] Kong W, Wei J, Abidi P, Lin M, Inaba S, Li C, Wang Y, Wang Z, Si S, Pan H, Wang S, Wu J, Wang Y, Li Z, Liu J, Jiang JD. Berberine is a novel cholesterol-lowering drug working through a unique mechanism distinct from statins. Nat Med. 2004 Dec;10(12):1344-51. doi: 10.1038/nm1135. Epub 2004 Nov 7. PMID 15531889
- [Background] Yuan X, Wang J, Tang X, Li Y, Xia P, Gao X. Berberine ameliorates nonalcoholic fatty liver disease by a global modulation of hepatic mRNA and lncRNA expression profiles. J Transl Med. 2015 Jan 27;13:24. doi: 10.1186/s12967-015-0383-6. PMID 25623289
- [Background] Zhang Z, Li B, Meng X, Yao S, Jin L, Yang J, Wang J, Zhang H, Zhang Z, Cai D, Zhang Y, Ning G. Berberine prevents progression from hepatic steatosis to steatohepatitis and fibrosis by reducing endoplasmic reticulum stress. Sci Rep. 2016 Feb 9;6:20848. doi: 10.1038/srep20848. PMID 26857750
- [Background] Cao Y, Pan Q, Cai W, Shen F, Chen GY, Xu LM, Fan JG. Modulation of Gut Microbiota by Berberine Improves Steatohepatitis in High-Fat Diet-Fed BALB/C Mice. Arch Iran Med. 2016 Mar;19(3):197-203. PMID 26923892
- [Background] Yan HM, Xia MF, Wang Y, Chang XX, Yao XZ, Rao SX, Zeng MS, Tu YF, Feng R, Jia WP, Liu J, Deng W, Jiang JD, Gao X. Efficacy of Berberine in Patients with Non-Alcoholic Fatty Liver Disease. PLoS One. 2015 Aug 7;10(8):e0134172. doi: 10.1371/journal.pone.0134172. eCollection 2015. PMID 26252777
- [Background] Chalasani NP, Sanyal AJ, Kowdley KV, Robuck PR, Hoofnagle J, Kleiner DE, Unalp A, Tonascia J; NASH CRN Research Group. Pioglitazone versus vitamin E versus placebo for the treatment of non-diabetic patients with non-alcoholic steatohepatitis: PIVENS trial design. Contemp Clin Trials. 2009 Jan;30(1):88-96. doi: 10.1016/j.cct.2008.09.003. Epub 2008 Sep 10. PMID 18804555
- [Background] Pickering TG, Hall JE, Appel LJ, Falkner BE, Graves JW, Hill MN, Jones DH, Kurtz T, Sheps SG, Roccella EJ; Council on High Blood Pressure Research Professional and Public Education Subcommittee, American Heart Association. Recommendations for blood pressure measurement in humans: an AHA scientific statement from the Council on High Blood Pressure Research Professional and Public Education Subcommittee. J Clin Hypertens (Greenwich). 2005 Feb;7(2):102-9. doi: 10.1111/j.1524-6175.2005.04377.x. No abstract available. PMID 15722655
- [Background] Kleiner DE, Brunt EM, Van Natta M, Behling C, Contos MJ, Cummings OW, Ferrell LD, Liu YC, Torbenson MS, Unalp-Arida A, Yeh M, McCullough AJ, Sanyal AJ; Nonalcoholic Steatohepatitis Clinical Research Network. Design and validation of a histological scoring system for nonalcoholic fatty liver disease. Hepatology. 2005 Jun;41(6):1313-21. doi: 10.1002/hep.20701. PMID 15915461